CLINICAL TRIAL: NCT02690662
Title: Influence of Hypocaloric Diet on Urinary Lithogenic Factors of Obese Patients With Kidney Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP 2015/04998-1
Record Dates: First submitted 2016-02-15; First posted 2016-02-24 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2016-10

CONDITIONS: Obesity; Kidney Stones
Keywords: Obesity; Kidney stones; Diet
MeSH Terms: conditions — Obesity; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obese with kidney stones (Experimental): Hypocaloric diet for 3 months
  Interventions: Behavioral: Hypocaloric diet

INTERVENTIONS:
Behavioral: Hypocaloric diet — recommendation of daily ingestion of 2500 ml of water and low-calorie diet of 16 Kcal/kg bw/day

SUMMARY:
The objective of this study is to evaluate the influence of low-calorie diet on serum and urinary metabolic parameters of obese adults with urinary calculi and lithogenic metabolic abnormalities.

DETAILED DESCRIPTION:
Objective: to evaluate the influence of low-calorie diet on serum and urinary metabolic parameters of obese adults with urinary calculi and lithogenic metabolic abnormalities.

Method: prospective study of 50 patients, aged over 18 years, with a body mass index above 30 kg/m2, urinary calculi and lithogenic metabolic abnormalities. Will be excluded from the study patients with psychiatric diagnoses other than depression, patients with inability to attend to clinical follow-up, patients with nephrocalcinosis, patients with urinary tract infection, patients with cystinuria and patients subjected to previous surgeries to treat obesity. Each patient will be evaluated monthly on the same day by urologist and nutritionist. On the first evaluation, will be done anamnesis, anthropometric measurements of weight, height, waist, bioimpedance and requested total serum calcium, phosphate, sodium, potassium, urea, creatinine, uric acid, and PTH, pH venous blood, urine tests type I, culture of urine and urine tests of calcium, oxalate, phosphate, sodium, potassium, citrate, magnesium, creatinine, uric acid, cystine and computed tomography for evaluation of urinary calculus. In the second evaluation, 30 days after, anthropometric measures will be repeated, bioimpedance and nutritional assessment will be made with recommendation of daily ingestion of 2500 ml of water and low-calorie diet of 16 Kcal/kg bw/day and requested total serum calcium, phosphate, sodium, potassium, urea, creatinine, uric acid, and PTH, pH venous blood, urine tests type I, culture of urine and urine tests of calcium, oxalate, phosphate, sodium, potassium, citrate, magnesium, creatinine, uric acid, cystine. Patients will be monitored monthly for 3 months with anthropometric measurements, bioimpedance and strengthening of nutritional recommendations. By the end of the third month, patients will be submitted to two series of serum and urine tests as before the diet. The results of serum and urine tests from the beginning of dietary treatment will be compared to those of the end of the treatment with Student T test. P<0.05 are considered significant.

ELIGIBILITY:
Inclusion Criteria:

* body mass index above 30 kg/m2 and urinary calculi on tomography and lithogenic metabolic abnormalities.

Exclusion Criteria:

* psychiatric diagnoses other than depression
* inability to attend to clinical follow-up
* nephrocalcinosis
* urinary tract infection
* cystinuria
* previous surgeries to treat obesity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Urinary lithogenic factors variation | 3 months
  serum and 24h urine test as before the diet.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Danilovic, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Condensed data will be available for consultation